## Psychological treatment of hypersexuality: a clinical trial with Acceptance and Commitment Therapy

ID: CIPI/21/003

Document date: 8th January 2021

IP: Francisco Montesinos, Ph.D.

Study Protocol and Statistical Analysis Plan

## **Study Protocol:**

- Objective: To study the efficacy of an abridged intervention aimed at increasing psychological flexibility and sexual impulse control in people with clinically significant hypersexuality.
- Design: Open clinical trial without control group
- Methods.

After being informed about the study, all patients giving written informed consent will be assessed to determine eligibility for study entry. Patients who meet eligibility requirements will receive psychological intervention consisting in an 8-session individual on line-delivered ACT-based treatment. The participants will be assessed through self-report instruments before and after treatment and at 3 months follow-up. Self-monitoring measures will be completed before every session.

Intervention protocol.

Session 1. Values clarification. Funeral exercise (Hayes et al., 2012). Garden metaphor (Hayes et al., 2012).

Session 2. Creative hopelessness. Sharing functional analysis with the client. Control in the problem, not the solution. Hungry tiger metaphor (Eifert & Forsyth, 2005). Chocolate Cake task (Hayes et al., 2012). Establishing valued commitments in the presence of craving or discomfort.

Session 3. Increasing awareness of physical sensations and consequences of avoidance behaviors. Training cognitive defusion and promoting self-as-context. Physicalizing Exercise (Hayes et al., 2012). The Soldiers in the Parade exercise (Hayes et al., 2012). Exposure to cravings and discomfort exercise. Learning to choose which train to take. Establishing new valued commitments.

Session 4. Increasing psychological flexibility: learning how to choose. Training cognitive defusion and promoting self-as-context. Body-scan exercise (Segal et al., 2015, p.67). Exposure to cravings and discomfort exercise. Establishing a commitment of reducing hypersexual behaviors.

Session 5. Listening to the messages from our mind. Shops Street metaphor (Wilson & Luciano, 2002, p.115). Leaves on a stream meditation (Hayes et al., 2012). Establishing a new commitment of reducing hypersexual behaviors.

Session 6. Deepening in body awareness. Taking care of "my garden". Training cognitive defusion and promoting self-as-context. Body-scan exercise (Segal et al., 2015). Physicalizing Exercise (Hayes et al., 2012). Differentiating between values, goals, committed actions and barriers in on valued areas. Establishing new commitments.

Session 7. Making peace with emotional pain. Training cognitive defusion and promoting self-as-context. Learning to choose opening to discomfort in order to live a fulfilling life. Exposure exercise to deep pain. Self-compassion exercise.

Session 8. Relapse prevention. Bycicle metaphor (Hayes et al., 2012). Identifying future risk situations. Exposure exercise to future risk situations. Renewing commitments.

## **Statistical Analysis Plan (SAP):**

The results will be analysed through non-parametric techniques (comparisons of pre, post and follow-up group means). Within-subject analyses will be performed. Non-overlap effect size measures will be used to estimate the magnitude of therapeutic change. The statistical approach of Jacobson and Truax (1991) will be used to estimate the clinical significance of the effect.